CLINICAL TRIAL: NCT01549691
Title: Assessment of Two Modes of Premedication in Surgery - PREMED Study
Brief Title: Reassessment of Premedication in Surgery
Acronym: PREMED
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PHRC 2011-20; 2011-002553-65 (EudraCT Number)
Record Dates: First submitted 2012-02-23; First posted 2012-03-09 (Estimated); Last update posted 2013-09-25 (Estimated); Status verified 2013-09

CONDITIONS: Anxiety
Keywords: Premedication; Benzodiazepine; Anti-anxiety agents; Anxiety; Surgery; Adult; Human
MeSH Terms: conditions — Anxiety Disorders | interventions — zopiclone; Alprazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- zopiclone (Experimental): zopiclone given before sleep, the day before surgery (placebo given at awakening the day of surgery)
  Interventions: Drug: Zopiclone
- alprazolam (Experimental): given at awakening, the day of surgery (placebo given before sleep, the day before surgery)
  Interventions: Drug: Alprazolam
- placebo (Placebo Comparator): Placebo given night before operation and the morning of operation
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Zopiclone — 7.5 mg before sleep, the evening before surgery
  Other Names: Imovane
  Arms: zopiclone
Drug: Alprazolam — 0.5 mg at awakening, the day of surgery
  Other Names: Xanax
  Arms: alprazolam
Drug: placebo — given night before surgery and at awakening, the day of surgery
  Arms: placebo

SUMMARY:
The purpose of this study is to test the level of anxiety in patients, the day before surgery (late afternoon) and immediately prior to surgery in 3 parallel groups of patients.

* one receiving placebo before going to sleep (before sleep), the day prior surgery and placebo when awakening (awakening), the day of surgery
* one receiving zopiclone (7.5 mg) before sleep and placebo at awakening
* one receiving placebo before sleep and alprazolam (0.5 mg)at awakening

double blind, randomized controlled study

DETAILED DESCRIPTION:
Eligibility:

* 18 to 65 years old
* elective surgery
* in-hospital preoperative night

Outcome measures:

* anxiety scales
* demographic data

ELIGIBILITY:
Inclusion Criteria:

* age 18-65 years old
* elective surgery
* in-hospital night before surgery

Exclusion Criteria:

* myasthenia gravis
* chronic intake of psychotropic drugs
* opiates intake
* severe obstructive sleep apnea
* intracranial hypertension
* morbid obesity
* myasthenia gravis
* acute severe medical disorder
* non health insurance coverage
* protected patients by law
* pregnancy
* non French speaking

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 455 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
anxiety scales | duration of the study : 12 hours (one evaluation on late afternoon the day before surgery and the second evaluation on arrival to operating room)
  * The day before surgery (late afternoon) : patient's self rating of anxiety and desire of information regarding upcoming surgery (Amsterdam patient anxiety and information scale, APAIS)
  * On arrival to the operating room : Recording of the level of declared anxiety (numeric scale similar to that corresponding of the "anxiety component of the APAIS scale)

SECONDARY OUTCOMES:
markers of stress | on arrival to operating room (one single recording)
  recording of actual (using the operating room monitor):
  * heart rate (at rest, supine)
  * systolic blood pressure (at rest, supine)

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Beydon, MD, Study Chair — University Hospital Angers (Dept of Anesthesia)
Locations (8):
- France (8):
  - Clinique Sévigné, Cesson, Brittany Region
  - Dept of Anesthesia, Hôpital Maison Blanche, Reims, Champagne
  - Centre Paul Papin, Angers, Maine et Loire
  - University Hospital, Angers, Maine et Loire
  - Clinique St Leonard, Trélazé, Maine et Loire
  - Dept of Anesthesia, Le Mans, Maine
  - Dept of Anesthesia, Hôpital Tenon, Paris, Île-de-France Region
  - Dept of Anesthesia, Hôpital Foch,, Suresnes, Île-de-France Region

REFERENCES:
- [Derived] Beydon L, Rouxel A, Camut N, Schinkel N, Malinovsky JM, Aveline C, Marret E, Bildea A, Dupoiron D, Liu N, Daniel V, Darsonval A, Chretien JM, Rault L, Bruna J, Alberti C. Sedative premedication before surgery--A multicentre randomized study versus placebo. Anaesth Crit Care Pain Med. 2015 Jun;34(3):165-71. doi: 10.1016/j.accpm.2015.01.005. Epub 2015 May 23. PMID 26004882